CLINICAL TRIAL: NCT05498181
Title: Angiotensin-Neprilysin Inhibition in Hemodialysis Initiation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Finnian McCausland, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P003592; R01DK129749 (NIH)
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Hemodialysis
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Intervention Model Description: Parallel group randomized trial of sacubitril/valsartan versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded (quadruple) and placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- sacubitril/valsartan (Experimental): Participants will take sacubitril/valsartan, beginning dose of 24/26mg twice daily, with titration to target dose of 97/103 mg twice daily over the first four weeks. Patients will remain on the maximally tolerated dose for the remaining 12 weeks (total on-drug period of 16 weeks) before stopping drug and being followed for a further two weeks (total study time of 18 weeks).
  Interventions: Drug: Sacubitril-valsartan
- placebo (Placebo Comparator): Participants will take equivalent placebo, beginning equivalent dose of 24/26mg twice daily, with titration to target equivalent dose of 97/103 mg twice daily over the first four weeks. Patients will remain on the maximally tolerated dose for the remaining 12 weeks (total on-drug period of 16 weeks) before stopping drug/placebo and being followed for a further two weeks (total study time of 18 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sacubitril-valsartan — sacubitril/valsartan
  Other Names: Entresto
  Arms: sacubitril/valsartan
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
This randomized placebo-controlled clinical trial will evaluate the effect of sacubitril/valsartan (compared with placebo) on echocardiographic measures of hypervolemia, preservation of residual renal function, and key safety parameters in incident hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years initiating HD (within 90 days of first HD session)
* Thrice-weekly HD
* Informed consent
* Hemodynamically Stable: Sitting pre-dialysis SBP ≥110 mmHg averaged over prior two weeks or at the baseline visit; no symptomatic hypotension in prior two weeks; no use of midodrine.
* Has not taken an ACEi for 36 hours prior to randomization

Exclusion Criteria:

* Anuria (daily urine volume <100 mL/day)
* Current or any use of sacubitril/valsartan within the past 30 days
* History of hypersensitivity or intolerance to any of the study drugs, including ARBs or sacubitril/valsartan
* Angioedema related to previous ACE inhibitor, ARB, or ARNI therapy
* Serum potassium >5.5 mEq/L at screening (pre-HD if already on HD)
* Acute coronary syndrome, stroke, TIA, major CV surgery, percutaneous coronary intervention or carotid angioplasty within one month
* Intended coronary or carotid revascularization within 4 months
* Implantation of a cardiac resynchronization therapy device (CRTD) within 3 months or intent to implant a CRTD
* History of heart transplant, or planned heart transplant, or with left ventricular assist device
* Planned renal transplant within 4 months
* Documented untreated ventricular arrhythmia with syncopal episodes within 3 months
* Symptomatic bradycardia or 2nd or 3rd degree heart block without a pacemaker
* Presence of hemodynamically significant valvular disease or hypertrophic cardiomyopathy or infiltrative cardiomyopathy including suspected or confirmed amyloid heart disease (amyloidosis)
* History of malignancy of any organ system within the past year (exceptions: squamous and basal cell carcinomas of the skin and carcinoma of the cervix in situ, or a malignancy that in the opinion of the investigator is considered cured with minimal risk of recurrence)
* Liver disease (e.g., acute hepatitis, chronic active hepatitis, cirrhosis with evidence of portal hypertension); Alanine aminotransferase (ALT) levels >2.0 times the upper limit of normal (ULN) or total bilirubin >1.5 times the ULN, unless consistent with Gilbert's disease
* Pregnant (positive hCG test) or lactating women
* Enrollment in another interventional trial
* Received an active investigational drug (including vaccines) other than a placebo agent, or used an investigational medical device within 12 weeks before Day 1/baseline
* Does not have capacity to consent (Folstein mini-mental score of 23 or less)
* Any condition that in the opinion of the investigator would make participation not in the best interest of the subject
* Women of child-bearing age, unless using two birth control methods. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of investigational drug and for 7 days off of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in left atrial volume index from baseline to 16 weeks | 16 weeks
  Primary Efficacy Outcome

SECONDARY OUTCOMES:
Change in IVC collapsibility index from baseline to 16 weeks | 16 weeks
  Secondary Efficacy Outcome
Change in pre-dialysis NTpro-BNP from baseline to 16 weeks | 16 weeks
  Secondary Efficacy Outcome
Change in eGFR from baseline to 16 weeks, assessed by 24-hour averaged urien urea and creatinine clearance | 16 weeks
  Secondary Efficacy Outcome
Adverse Events frequency | 18 weeks (includes 2 weeks period off-treatment period)
  Safety Outcome
Serious Adverse Events frequency | 18 weeks (includes 2 weeks period off-treatment period)
  Safety Outcome
Inter-dialytic hypotension (symptomatic SBP <90 mmHg or hypotension requiring adjustment in blood pressure medications or treatment in an emergency or hospitalized setting) frequency | 18 weeks (includes 2 weeks period off-treatment period)
  Safety Outcome
Intra-dialytic hypotension (defined as nadir SBP <90 mmHg if pre-HD SBP≤160 mmHg, or nadir SBP <100 mmHg if pre-HD SBP >160 mmHg) frequency | 18 weeks (includes 2 weeks period off-treatment period)
  Safety Outcome
Hyperkalemia (pre-dialysis serum potassium >5.5 mmol/L) frequency | 18 weeks (includes 2 weeks period off-treatment period)
  Safety Outcome
Angioedema frequency | 18 weeks (includes 2 weeks period off-treatment period)
  Safety Outcome
Proportion of participants able to complete the full 16 weeks of treatment | 16 weeks
  Tolerability Outcome
Proportion of participants able to reach maximum dose titration | 16 weeks
  Tolerability Outcome
Study medication discontinuation rates | 16 weeks
  Tolerability Outcome
Changes in SMaRRT-HD and Dialysis Symptom Index questionnaire scores from baseline to 16 weeks | 16 weeks
  Tolerability Outcome
Rates of recruitment, withdrawal, and loss-to-follow-up | 18 weeks
  Tolerability Outcome
Reasons for ineligibility | Baseline
  Tolerability Outcome
Adherence to the study drug administration schedule | 16 weeks
  Tolerability Outcome

OTHER OUTCOMES:
Change in pre-HD hsTnT from baseline to 16 weeks | 16 weeks
  Exploratory Outcome
Heart failure hospitalization/ hospitalization with volume overload frequency | 18 weeks
  Exploratory Outcome
All-cause mortality | 18 weeks
  Exploratory Outcome
Death from cardiovascular causes | 18 weeks
  Exploratory Outcome

CONTACTS AND LOCATIONS:
Overall Officials: Finnian Mc Causland, MBBCh, MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Only sharing of anonymized data will be considered as per approved protocol. Written requests for data sharing will be considered on a case-by-case basis from qualified external researchers, based on scientific merit.

REFERENCES:
- [Background] Solomon SD, McMurray JJV, Anand IS, Ge J, Lam CSP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rouleau JL, van Veldhuisen DJ, Zannad F, Zile MR, Desai AS, Claggett B, Jhund PS, Boytsov SA, Comin-Colet J, Cleland J, Dungen HD, Goncalvesova E, Katova T, Kerr Saraiva JF, Lelonek M, Merkely B, Senni M, Shah SJ, Zhou J, Rizkala AR, Gong J, Shi VC, Lefkowitz MP; PARAGON-HF Investigators and Committees. Angiotensin-Neprilysin Inhibition in Heart Failure with Preserved Ejection Fraction. N Engl J Med. 2019 Oct 24;381(17):1609-1620. doi: 10.1056/NEJMoa1908655. Epub 2019 Sep 1. PMID 31475794
- [Background] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Background] Mc Causland FR, Lefkowitz MP, Claggett B, Anavekar NS, Senni M, Gori M, Jhund PS, McGrath MM, Packer M, Shi V, Van Veldhuisen DJ, Zannad F, Comin-Colet J, Pfeffer MA, McMurray JJV, Solomon SD. Angiotensin-Neprilysin Inhibition and Renal Outcomes in Heart Failure With Preserved Ejection Fraction. Circulation. 2020 Sep 29;142(13):1236-1245. doi: 10.1161/CIRCULATIONAHA.120.047643. Epub 2020 Aug 17. PMID 32845715